CLINICAL TRIAL: NCT04053764
Title: A Phase II, Multicenter, Randomized, Open Label Two Arm Study Evaluating the Effect of Crizanlizumab + Standard of Care and Standard of Care Alone on Renal Function in Sickle Cell Disease Patients ≥ 16 Years With Chronic Kidney Disease Due to Sickle Cell Nephropathy (STEADFAST)
Brief Title: Study Exploring the Effect of Crizanlizumab on Kidney Function in Patients With Chronic Kidney Disease Caused by Sickle Cell Disease
Acronym: STEADFAST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSEG101A2203; 2018-003608-38 (EudraCT Number)
Record Dates: First submitted 2019-08-09; First posted 2019-08-12 (Actual); Results first posted 2024-06-04 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Sickle Cell Disease (SCD)
Keywords: SEG101; Sickle Cell Disease; SCD; Crizanlizumab; Sickle cell nephropathy; chronic kidney disease; CKD; albuminuria (ACR); renal function; standard of care
MeSH Terms: conditions — Anemia, Sickle Cell; Renal Insufficiency, Chronic; Albuminuria | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- crizanlizumab + standard of care (Experimental): 5 mg/kg by intravenous (i.v.) infusion at Week 1 Day 1, Week 3 Day 1 and Day 1 of every 4-week cycle until Week 51 in addition to their usual standard of care treatment.
  Interventions: Drug: Crizanlizuamb; Drug: Standard of Care
- standard of care (Active Comparator): Patients in the standard of care alone arm will continue to receive their usual standard of care treatment.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Crizanlizuamb — Crizanlizumab is a concentrate for solution for infusion, i.v. use. Supplied in single use 10 mL vials at a concentration of 10 mg/mL. One vial contains 100 mg of crizanlizumab
  Other Names: SEG101
  Arms: crizanlizumab + standard of care
Drug: Standard of Care — HU/HC (hydroxyurea/hydroxycarbamide) and/or ACE (angiotensin-converting enzyme) inhibitors and/or ARBs (angiotensin-receptor blocker)

SUMMARY:
The goal of the study was to evaluate descriptively the effect of crizanlizumab + standard of care and standard of care alone on renal function in sickle cell disease patients ≥ 16 years with chronic kidney disease due to sickle cell nephropathy.

DETAILED DESCRIPTION:
Approximately 50 patients were to be randomized 1:1 to receive either crizanlizumab (5 mg/kg) + standard of care or standard of care alone. Patients were stratified at randomization based on chronic kidney disease (CKD) risk category (moderate risk or high/very high risk) and hydroxyurea/hydroxycarbamide (HU/HC) prescription (Yes/No). The CKD risk categories used for stratification were based on both Estimated glomerular filtration rate(eGFR) and albuminuria assessed by Albumin/creatinine ratio (ACR).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of SCD (HbSS and HbSβ0-thal SCD genotypes are eligible)
* Patients with eGFR ≥ 45 to ≤ 140 mL/min/1.73 m2 based on CKD EPI formula (patients ≥ 18) or the Creatinine-based "Bedside Schwartz" equation (patients < 18)
* Patients with ACR of ≥ 100 to < 2000 mg/g (taken as an average of the three screening ACR values to determine eligibility)
* Receiving at least 1 standard of care drug(s) for SCD-related CKD: If receiving HU/HC, the patient must have been receiving HU/HC for at least 6 months and on a stable dose for 3 months, and/or an ACE inhibitor and/or ARB for 3 months and on a stable dose for those 3 months.
* Hb ≥ 4.0 g/dL, absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L, and platelet count ≥ 75 x 10^9/L
* Adequate hepatic function as defined by:

  * Alanine aminotransferase (ALT) < 3.0 x upper limit of normal (ULN)
  * Direct (conjugated) bilirubin ≤ 3.0 x ULN
* Written informed consent (or assent/ parental consent for minor subjects) prior to any screening procedures

Exclusion Criteria:

* History of stem cell transplant
* Patients with evidence of AKI within 3 months of study entry (can decrease interval to within 6 weeks of study entry only if renal function has returned to pre-AKI values prior to study entry)
* Blood pressure > 140/90 mmHg despite treatment
* Patients undergoing renal replacement therapy (ie. hemodialysis, peritoneal dialysis, hemofiltration and kidney transplantation)
* Received blood products within 30 days of Week 1 Day 1
* Participating in a chronic transfusion program
* History of kidney transplant
* Patients with hypoalbuminemia
* Body mass index of ≥ 35
* Currently receiving or received voxelotor within 6 months of screening
* Patient has received crizanlizumab and/or other selectin inhibitor or plans to receive it during the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- United States (6):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of Illinois Hospital and Health Sciences System ., Chicago, Illinois
  - Our Lady of the Lake Regional Medic ., Baton Rouge, Louisiana
  - East Carolina University BrodySchool of Med 3, Greenville, North Carolina
  - Univ of Tenn Health Sciences Ctr, Memphis, Tennessee
  - University of Texas Health Science Center at Houston, Houston, Texas
- Brazil (3):
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Porto Alegre
- France (2):
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Paris
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Larissa
- Novartis Investigative Site, Dublin, Ireland
- Novartis Investigative Site, Tripoli, Lebanon
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, Panama City, Panama
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Antakya / Hatay
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Abbasi M, Srivastava A, Saraf SL. Management of Kidney Disease with Sickle Cell Disease. J Am Soc Nephrol. 2025 Oct 1;36(10):2041-2054. doi: 10.1681/ASN.0000000804. Epub 2025 Jun 26. PMID 40569673
- [Derived] Obadina M, Wilson S, Derebail VK, Little J. Emerging Therapies and Advances in Sickle Cell Disease with a Focus on Renal Manifestations. Kidney360. 2023 Jul 1;4(7):997-1005. doi: 10.34067/KID.0000000000000162. Epub 2023 May 31. PMID 37254256
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled in 24 centers in 11 countries.
Pre-assignment Details: Patients were stratified at randomization based on CKD risk category (moderate risk or high/very high risk) and HU/HC use (Yes/No).
  At visit "Week 1 Day 1" all eligible patients were randomized via Interactive Response Technology (IRT) to one of the treatment arms.
Groups:
- Standard of Care (SOC): Patients in the standard of care alone arm will continue to receive their usual standard of care treatment.
Period: Overall Study
Arm/Group | Crizanlizumab + Standard of Care | Standard of Care (SOC)
Started | 30 | 28
Entered Post-treatment Follow-up, Discontinued | 7 | 1
Did Not Enter Post-treatment Follow-up | 3 | 2
Not Treated | 1 | 0
Completed (Completed = completed treatment Not Completed = discontinued treatment) | 20 | 25
Not Completed | 10 | 3
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Physician Decision | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Pregnancy | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Crizanlizumab + Standard of Care | Standard of Care (SOC) | Total
Number analyzed (Participants) | 30 | 28 | 58
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.8 (9.52) | 41.1 (8.71) | 41.5 (9.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 10 | 11 | 21
Race/Ethnicity, Customized [Number; unit: Participants] — Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
  Participants
    Black or African American | 15 | 15 | 30
    White | 15 | 12 | 27
    Multiple | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ≥ 30% Decrease in Albuminuria (ACR) at 12 Months
Description: The effect of SEG101 on clinical disease activity was measured by at least 30% decrease in Albumin to Creatinine Ratio (ACR) from baseline to month 12. A reduction from baseline indicates improvement in patients.
Time Frame: Baseline to 12 months
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | Crizanlizumab + Standard of Care | Standard of Care (SOC)
Number analyzed (Participants) | 30 | 28
Percentage of participants | 33.3 | 21.4
Statistical Analysis 1: Comparison: Crizanlizumab + Standard of Care vs Standard of Care (SOC); Test type: Superiority; Odds Ratio (OR) = 1.94, 95% CI 2-sided [0.53 to 7.14]

2. Secondary Outcome: Change From Baseline in Albuminuria (ACR) at 3, 6, 9 and 12 Months
Description: The effect of SEG101 on clinical disease activity was measured by the change in albuminuria (ACR) between baseline and month 3, baseline and month 6, baseline and month 9, baseline and month 12. A reduction from baseline indicates improvement in patients.
Time Frame: Baseline to 3, 6, 9, and 12 months
Population: Participants in the FAS with an available assessment for the outcome measure at baseline and at each timepoint. The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Crizanlizumab + Standard of Care | Standard of Care (SOC)
Number analyzed (Participants) | 29 | 28
mg/g
  Baseline (BL) | 597.0 (534.3) | 499.0 (486.7)
  Month 3 change from BL: number analyzed (Participants) | 26 | 27
  Month 3 change from BL | -56.9 (362.8) | 159.0 (809.9)
  Month 6 change from BL: number analyzed (Participants) | 23 | 25
  Month 6 change from BL | -98.5 (382.2) | -35.4 (384.4)
  Month 9 change from BL: number analyzed (Participants) | 23 | 24
  Month 9 change from BL | -12.3 (586.6) | 95.2 (376.2)
  Month 12 change from BL: number analyzed (Participants) | 21 | 24
  Month 12 change from BL | 17.7 (620.7) | 14.7 (307.1)

3. Secondary Outcome: Percentage of Participants With ≥ 30% Decrease in Albuminuria (ACR) at 6 Months
Description: The effect of SEG101 on clinical disease activity was measured by at least 30% decrease in Albumin to Creatinine Ratio (ACR) from baseline to month 6. A reduction from baseline indicates improvement in patients.
Time Frame: Baseline to 6 months
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | Crizanlizumab + Standard of Care | Standard of Care (SOC)
Number analyzed (Participants) | 30 | 28
Percentage of participants | 30.0 | 35.7
Statistical Analysis 1: Comparison: Crizanlizumab + Standard of Care vs Standard of Care (SOC); Test type: Superiority; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.23 to 2.31]

4. Secondary Outcome: Percentage of Participants With Protein/Creatinine Ratio (PCR) Improvement and Stable PCR at 12 Months
Description: The effect of SEG101 on clinical disease activity was measured by counting patients who had Stable PCR: within ± 20% change from baseline to month 12. PCR improvement: ≥ 20% decrease in PCR from baseline indicates improvement in patients.
Time Frame: Baseline to 12 months
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | Crizanlizumab + Standard of Care | Standard of Care (SOC)
Number analyzed (Participants) | 30 | 28
Percentage of participants
  Percentage of participants with PCR improvement at 12 months | 33.3 | 35.7
  Percentage of participants with stable PCR at 12 months | 16.7 | 25.0
Statistical Analysis 1: Comparison: Crizanlizumab + Standard of Care vs Standard of Care (SOC); PCR Improvement; Test type: Superiority; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.29 to 3.02]
Statistical Analysis 2: Comparison: Crizanlizumab + Standard of Care vs Standard of Care (SOC); Stable PCR; Test type: Superiority; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.18 to 3.20]

5. Secondary Outcome: Percentage Change From Baseline in Estimated Glomerular Filtration Rate (eGFR)
Description: The percentage change in eGFR was calculated as the post-baseline eGFR value minus the baseline eGFR divided by the eGFR at baseline. A reduction from baseline indicates improvement in participants.
Time Frame: Baseline to 3, 6, 9, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage change in eGFR
Arm/Group | Crizanlizumab + Standard of Care | Standard of Care (SOC)
Number analyzed (Participants) | 28 | 28
Percentage change in eGFR
  Month 3 change from BL: number analyzed (Participants) | 24 | 26
  Month 3 change from BL | -2.5 (8.9) | -0.5 (10.0)
  Month 6 change from BL: number analyzed (Participants) | 21 | 25
  Month 6 change from BL | -2.7 (5.5) | -7.3 (12.7)
  Month 9 change from BL: number analyzed (Participants) | 23 | 23
  Month 9 change from BL | -0.2 (12.8) | -2.7 (8.7)
  Month 12 change from BL: number analyzed (Participants) | 16 | 24
  Month 12 change from BL | -4.9 (14.1) | -6.3 (13.2)
Statistical Analysis 1: Comparison: Crizanlizumab + Standard of Care vs Standard of Care (SOC); From baseline to 3 months; Test type: Superiority; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-5.53 to 4.65], Standard Error of Mean 2.53
Statistical Analysis 2: Comparison: Crizanlizumab + Standard of Care vs Standard of Care (SOC); From baseline to 6 months; Test type: Superiority; Mean Difference (Final Values) = 4.69, 95% CI 2-sided [-2.02 to 11.40], Standard Error of Mean 3.32
Statistical Analysis 3: Comparison: Crizanlizumab + Standard of Care vs Standard of Care (SOC); From baseline to 9 months; Test type: Superiority; Mean Difference (Final Values) = 4.05, 95% CI 2-sided [-3.58 to 11.68], Standard Error of Mean 3.77
Statistical Analysis 4: Comparison: Crizanlizumab + Standard of Care vs Standard of Care (SOC); From baseline to 12 months; Test type: Superiority; Mean Difference (Final Values) = 5.19, 95% CI 2-sided [-3.28 to 13.67], Standard Error of Mean 4.17

6. Secondary Outcome: Slope of Albumin to Creatinine Ratio (ACR) Decline
Description: The effect of SEG101 on clinical disease activity was measured by the slope of ACR decline between baseline and Month 12. A reduction from baseline indicates improvement in patients.
Time Frame: Baseline to 12 months
Population: Participants in the FAS with an available assessment for the outcome measure at baseline and up to 12 months. The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
Measure: Least Squares Mean (Standard Error); unit: mg/g per month
Arm/Group | Crizanlizumab + Standard of Care | Standard of Care (SOC)
Number analyzed (Participants) | 29 | 28
mg/g per month | 1.70 (8.655) | 4.49 (8.159)

7. Secondary Outcome: Slope of Estimated Glomerular Filtration Rate (eGFR) Decline
Description: The effect of SEG101 on clinical disease activity was measured by the slope of eGFR between baseline and Month 12. The calculation of eGFR is based on the chronic kidney disease epidemiology collaboration (CKD-EPI) (for patients ≥ 18) and Creatinine-based "Bedside Schwartz" (for patients < 18) equations. A reduction in drop rate from baseline indicates improvement in patients.
Time Frame: Baseline to 12 months
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2 per month
Arm/Group | Crizanlizumab + Standard of Care | Standard of Care (SOC)
Number analyzed (Participants) | 28 | 28
mL/min/1.73 m^2 per month | -0.1 (0.18) | -0.4 (0.16)

8. Secondary Outcome: Percentage of Participants With Progression of Chronic Kidney Disease (CKD) at 12 Months
Description: The effect of SEG101 on clinical disease activity was measured by percentage of participants with CKD progression between baseline and Month 12. A reduction from baseline indicates improvement in participants.
  CKD progression is defined as an increase in CKD progression category, a 25% or greater drop in eGFR from baseline or at least 50% increase in ACR for patients with severe (A3) albuminuria and a doubling of albumin levels in patients with moderate (A2) albuminuria.
Time Frame: Baseline to 12 months
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | Crizanlizumab + Standard of Care | Standard of Care (SOC)
Number analyzed (Participants) | 30 | 28
Percentage of participants | 13.3 | 32.1
Statistical Analysis 1: Comparison: Crizanlizumab + Standard of Care vs Standard of Care (SOC); Test type: Superiority; Odds Ratio (OR) = 0.32, 95% CI 2-sided [0.09 to 1.21]

9. Secondary Outcome: Shift Table for Chronic Kidney Disease (CKD) Progression
Description: The effect of SEG101 on clinical disease activity was measured by percentage of participants with CKD progression between baseline and Month 12. A reduction from baseline indicates improvement in patients.
Time Frame: Baseline and month 12
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
Measure: Number; unit: Percentage of participants
Groups:
- All Patients: All the participants enrolled in the trial.
Arm/Group | Crizanlizumab + Standard of Care | Standard of Care (SOC) | All Patients
Number analyzed (Participants) | 30 | 28 | 58
Percentage of participants
  Cat 0 at baseline | 3.3 | 14.3 | 8.6
  Cat 0 at baseline to Cat 2 at Worst post-baseline | 100.0 | 75.0 | 80.0
  Cat 0 at baseline to Cat 3 at Worst post-baseline | 0 | 25.0 | 20.0
  Cat 0 at baseline to Cat 4 at Worst post-baseline | 0 | 0 | 0
  Cat 0 at baseline to Missing at Worst post-baseline | 0 | 0 | 0
  Cat 1 at baseline | 36.7 | 53.6 | 44.8
  Cat 1 at baseline to Cat 2 at Worst post-baseline | 36.4 | 40.0 | 38.5
  Cat 1 at baseline to Cat 3 at Worst post-baseline | 45.5 | 53.3 | 50.0
  Cat 1 at baseline to Cat 4 at Worst post-baseline | 0 | 6.7 | 3.8
  Cat 1 at baseline to Missing at Worst post-baseline | 18.2 | 0 | 7.7
  Cat 2 at baseline | 43.3 | 28.6 | 36.2
  Cat 2 at baseline to Cat 2 at Worst post-baseline | 15.4 | 12.5 | 14.3
  Cat 2 at baseline to Cat 3 at Worst post-baseline | 69.2 | 75.5 | 71.4
  Cat 2 at baseline to Cat 4 at Worst post-baseline | 7.7 | 12.5 | 9.5
  Cat 2 at baseline to Missing at Worst post-baseline | 7.7 | 0 | 4.8
  Cat 3 at baseline | 6.7 | 3.6 | 5.2
  Cat 3 at baseline to Cat 2 at Worst post-baseline | 0 | 0 | 0
  Cat 3 at baseline to Cat 3 at Worst post-baseline | 50.0 | 0 | 33.3
  Cat 3 at baseline to Cat 4 at Worst post-baseline | 50.0 | 100.0 | 66.7
  Cat 3 at baseline to Missing at Worst post-baseline | 0 | 0 | 0
  Cat 4 at baseline | 0 | 0 | 0
  Cat 4 at baseline to Cat 2 at Worst post-baseline | 0 | 0 | 0
  Cat 4 at baseline to Cat 3 at Worst post-baseline | 0 | 0 | 0
  Cat 4 at baseline to Cat 4 at Worst post-baseline | 0 | 0 | 0
  Cat 4 at baseline to Missing at Worst post-baseline | 0 | 0 | 0
  Cat Missing at baseline | 10.0 | 0 | 5.2
  Cat Missing baseline to Cat 2 at Worst post-baseline | 0 | 0 | 0
  Cat Missing baseline to Cat 3 at Worst post-baseline | 0 | 0 | 0
  Cat Missing baseline to Cat 4 at Worst post-baseline | 0 | 0 | 0
  Cat Missing baseline to Missing at Worst post-baseline | 100.0 | 0 | 100.0

10. Secondary Outcome: Immunogenicity: Percentage of Participants With Anti-drug Antibodies (ADA) to Crizanlizumab
Description: The effect of SEG101 on clinical disease activity was measured by percentage of participants shifted to different worst post-baseline categories between baseline and Month 12. An increase in percentage shifting from higher category to lower category indicates improvement in patients.
  Baseline is defined as the last non-missing value prior to the first dose.
Time Frame: Baseline to follow-up period (at select time points), assessed up to approximately 1 year and 4 months
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Crizanlizumab + Standard of Care
Number analyzed (Participants) | 29
Percentage of participants
  Negative at baseline to Only last sample positive | 0
  Negative at baseline to Any positive | 3.4
  Negative at baseline to All positive | 0
  Negative at baseline to All Negative | 89.7
  Negative at baseline to All Missing | 6.9

11. Secondary Outcome: Annualized Rate of Visits to Emergency Room (ER) and Hospitalizations
Description: The effect of SEG101 on clinical disease activity was measured by summarizing the annualized rate of visits to ER and hospitalizations between baseline and 1 year 4 months. Annualized rate of hospitalizations and ER visits due to VOC =(Number of ER or hospitalizations reported until End date x 365.25)/(End date-date of first dose of study treatment+1). A reduction from baseline indicates improvement in patients.
Time Frame: Baseline to follow-up period (at select time points), assessed up to approximately 1 year and 4 months
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
Measure: Mean (Standard Deviation); unit: ER or hospitalizations/year
Arm/Group | Crizanlizumab + Standard of Care | Standard of Care (SOC)
Number analyzed (Participants) | 30 | 28
ER or hospitalizations/year | 0.6 (2.1) | 1.1 (3.0)

12. Secondary Outcome: Mean Serum Concentration (Ctrough) of Crizanlizumab
Description: The effect of SEG101 on clinical disease activity was measured by checking the concentration of the Drug in serum at different time points.
  Crizanlizumab pre-dose/trough pharmacokinetic samples were taken at select time points.
Time Frame: Pre-dose and 336 hours post-dose on Week 3 Day 1; pre-dose and 672 hours post dose on Week 11 Day 1, Week 23 Day 1 and Week 39 Day 1; and 672 hours post dose on Week 53 Day 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Crizanlizumab + Standard of Care
Number analyzed (Participants) | 29
μg/mL
  Week 3 Day1: 0 hours pre-dose: number analyzed (Participants) | 25
  Week 3 Day1: 0 hours pre-dose | 11.6 (2.66)
  Week 3 Day1: 336 hours post-dose: number analyzed (Participants) | 24
  Week 3 Day1: 336 hours post-dose | 12.1 (2.38)
  Week 11 Day1: 0 hours pre-dose: number analyzed (Participants) | 24
  Week 11 Day1: 0 hours pre-dose | 4.78 (3.49)
  Week 11 Day1: 672 hours post-dose: number analyzed (Participants) | 23
  Week 11 Day1: 672 hours post-dose | 5.67 (3.11)
  Week 23 Day1: 0 hours pre-dose: number analyzed (Participants) | 23
  Week 23 Day1: 0 hours pre-dose | 4.77 (2.82)
  Week 23 Day1: 672 hours post-dose: number analyzed (Participants) | 21
  Week 23 Day1: 672 hours post-dose | 5.54 (2.21)
  Week 39 Day1: 0 hours pre-dose: number analyzed (Participants) | 20
  Week 39 Day1: 0 hours pre-dose | 5.55 (2.34)
  Week 39 Day1: 672 hours post-dose: number analyzed (Participants) | 17
  Week 39 Day1: 672 hours post-dose | 5.16 (2.10)
  Week 53 Day1: 672 hours post-dose: number analyzed (Participants) | 16
  Week 53 Day1: 672 hours post-dose | 15.2 (5.18)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from first dose of study treatment to 105 days after the last dose of study treatment with a median duration of exposure to crizanlizumab of 50.1 weeks.
Description: Any sign or symptom that occurs during conduct of the trial & safety follow-up. Other AE: AE that is not an SAE, meaning it does not result in death, is not life-threatening, does not require inpatient hospitalization or extend a current hospital stay, does not result in an ongoing or significant incapacity, or interfere substantially with normal life functions & does not cause a congenital anomaly or birth defect. 1 subject randomized to the Crizanlizumab + Standard of Care arm was not treated.
Groups:
- All Participants: All Participants enrolled in the trial from whom safety was collected.
Arm/Group | Crizanlizumab + Standard of Care | Standard of Care (SOC) | All Participants
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28 | 0/57
Serious Adverse Events (participants affected / at risk) | 2/29 | 2/28 | 4/57
Other Adverse Events (participants affected / at risk) | 21/29 | 19/28 | 40/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crizanlizumab + Standard of Care (N=29) | Standard of Care (SOC) (N=28) | All Participants (N=57)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 | 1 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 1
Influenza (Infections and infestations) | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Crizanlizumab + Standard of Care (N=29) | Standard of Care (SOC) (N=28) | All Participants (N=57)
Tachycardia (Cardiac disorders) | 0 | 2 | 2
Constipation (Gastrointestinal disorders) | 3 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 2
Nausea (Gastrointestinal disorders) | 4 | 5 | 9
Vomiting (Gastrointestinal disorders) | 1 | 7 | 8
Fatigue (General disorders) | 2 | 3 | 5
Oedema peripheral (General disorders) | 0 | 3 | 3
Pyrexia (General disorders) | 3 | 2 | 5
COVID-19 (Infections and infestations) | 7 | 4 | 11
Influenza (Infections and infestations) | 4 | 4 | 8
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 2
Pharyngitis (Infections and infestations) | 2 | 1 | 3
Subcutaneous abscess (Infections and infestations) | 2 | 0 | 2
Tooth infection (Infections and infestations) | 4 | 0 | 4
Urinary tract infection (Infections and infestations) | 3 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 6
Headache (Nervous system disorders) | 6 | 4 | 10
Migraine (Nervous system disorders) | 2 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e., data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT04053764/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/64/NCT04053764/SAP_001.pdf